CLINICAL TRIAL: NCT00849628
Title: Use of Drugs and Constipation in Nursing Homes
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Other Study IDs: SI 150069-1
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Constipation; Diarrhea
Keywords: Aged; Polypharmacy; Adverse effects; Nursing homes
MeSH Terms: conditions — Constipation; Diarrhea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Constipation

SUMMARY:
The purpose of this study is to study factors (drugs, serum concentration of drugs, nutrition, physical activity, demographics, diseases etc.) related to constipation and diarrhea in nursing homes, and the effect of different laxative regimens.

ELIGIBILITY:
Inclusion Criteria:

* Above 60 years old
* Stayed in nursing homes for more than 8 weeks
* Informed consent

Exclusion Criteria:

* Expected discharge within 2 weeks
* Organic disorders causing constipation and diarrhea

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents in nursing homes
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of constipation | One year

CONTACTS AND LOCATIONS:
Overall Officials: Per G Farup, PhD, Principal Investigator — Sykehuset Innlandet HF
Locations (1):
- Innlandet Hospital Trust, Gjøvik, Oppland, Norway

REFERENCES:
- [Result] Fosnes GS, Lydersen S, Farup PG. Drugs and constipation in elderly in nursing homes: what is the relation? Gastroenterol Res Pract. 2012;2012:290231. doi: 10.1155/2012/290231. Epub 2012 Feb 29. PMID 22505881